CLINICAL TRIAL: NCT07163572
Title: Safety and Efficacy of Intravenous Brivaracetam Versus Levetiracetam in the Management of Status Epilepticus in Children
Brief Title: Comparison of Intravenous Brivaracetam Versus Levetiracetam in the Management of Status Epilepticus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dr-Ikram-Multan
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Status Epilepticus
MeSH Terms: conditions — Status Epilepticus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brivaracetam group (Experimental): Patients received brivaracetam as a loading dose of 2 mg/kg (maximum 100 mg) diluted in 100 ml of normal saline infused over 10 minutes.
  Interventions: Drug: Intravenous brivaracetam
- Levetiracetam group (Experimental): Patients received levetiracetam as a loading dose of 40 mg/kg (maximum 3000 mg) diluted in 100 ml of normal saline infused over 10 minutes.
  Interventions: Drug: Intravenous levetiracetam

INTERVENTIONS:
Drug: Intravenous brivaracetam — Patients received intravenous brivaracetam as a loading dose of 2 mg/kg (maximum 100 mg) diluted in 100 ml of normal saline infused over 10 minutes.
  Arms: Brivaracetam group
Drug: Intravenous levetiracetam — Patients received intravenous levetiracetam as a loading dose of 40 mg/kg (maximum 3000 mg) diluted in 100 ml of normal saline infused over 10 minutes.
  Arms: Levetiracetam group

SUMMARY:
Brivaracetam is increasingly being studied in adult status epilepticus populations, evidence in pediatric patients remains sparse, with only limited case series and observational studies reporting favorable outcomes. This study aims at direct comparison between intravenous brivaracetam and levetiracetam in the acute management of pediatric status epilepticus.

DETAILED DESCRIPTION:
Given the urgent need for safe and effective alternatives in pediatric status epilepticus and the limited head-to-head data comparing intravenous brivaracetam with levetiracetam, especially in children, this study has been designed to evaluate their relative safety and efficacy. The research seeks to generate evidence that may help guide clinical decision-making and optimize outcomes in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Either gender
* Aged one month to 16 years
* Presenting with status epilepticus

Exclusion Criteria:

* Previously received intravenous antiseizure medication for the current episode prior to presentation
* Known hypersensitivity to study drugs
* Hemodynamically unstable, requiring inotropic support before administration

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 152 (Actual)
Dates: Start 2025-01-16 (Actual); Primary Completion 2025-08-16 (Actual); Study Completion 2025-08-16 (Actual)

PRIMARY OUTCOMES:
Cessation of seizures | 30 minutes
  Cessation of seizures was labeled "yes" if cessation of clinical seizures occurred within 20-30 minutes of infusion without the need for additional antiseizure medication.

SECONDARY OUTCOMES:
Adverse Events | 40 minutes
  Labeled "yes" if any treatment-related adverse event reported 30 minutes post-infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Ikram Rahman, Principal Investigator — Children's Hospital and institute of Child Health, Multan, Pakistan; Nuzhat Noureen, FCPS, Study Director — Children's Hospital and institute of Child Health, Multan, Pakistan
Locations (1):
- The Children's Hospital and Institute of Child Health, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.